CLINICAL TRIAL: NCT03998852
Title: In Vivo Involvement of the Cholinergic and Dopaminergic Systems in the Pathophysiology of Apathy.
Acronym: ADACHOL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2017/22
Record Dates: First submitted 2019-06-20; First posted 2019-06-26 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Apathy
Keywords: Apathy; Stroke; Cholinergic neurotransmission; Dopaminergic neurotransmission
MeSH Terms: conditions — Lethargy; Stroke | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; fluorodopa F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Molecular imaging (Experimental): Positron Emission Tomography (PET) molecular imaging of dopaminergic and cholinergic systems using two radiotracers
  Interventions: Drug: Positron Emission Tomography (PET) with [18F]-FDOPA; Drug: Positron Emission Tomography (PET) with [18F]-FEOBV; Device: Magnetic Resonnance Imaging (MRI); Other: Neuropsychological evaluation

INTERVENTIONS:
Drug: Positron Emission Tomography (PET) with [18F]-FDOPA — Positron Emission Tomography (PET) with [18F]-FDOPA
Drug: Positron Emission Tomography (PET) with [18F]-FEOBV — Positron Emission Tomography (PET) with [18F]-FEOBV
Device: Magnetic Resonnance Imaging (MRI) — MRI protocol will be performed on the same day that the [18F]-FEOBV PET imaging, using a 3T scanner (Philips Medical System). Different types of images will be acquired.
Other: Neuropsychological evaluation — Neuropsychological evaluation will be performed, consisting in an assessment of apathy by actigraphy (social or physical activities will be recorded during seven days) and a complementary assessment of apathy using the Lille Apathy Rating Scale (LARS)

SUMMARY:
Apathy is a neurocognitive syndrome characterized by reduced goal-directed behaviors, contributing to decreased patient and caregiver quality of life. Apathy pathophysiology involves disruption of cortico-striato-thalamo-cortical loops, modulated by several neurotransmitter systems including dopamine and acetylcholine, thus complexifying pharmacological management. Post-stroke apathy (PSA) can provide a proper in vivo model to study the underlying neurochemical substrates of apathy as a syndrome. The present project aims to provide a better characterization of the cholinergic and dopaminergic functioning in apathy as a syndrome.

In order to precise the respective alterations of these two systems, investigators will use a positron emission tomography (PET) molecular imaging of dopaminergic (with [18F]-FDOPA, a marker of the decarboxylating enzyme of dopamine) and - for the first time in apathetic patients - cholinergic (with [18F]-FEOBV, a marker of the vesicular acetylcholine transporter) transmissions in 15 apathetic and 15 unapathetic patients 3 months after stroke, without overlapping depression. This dual imaging study may provide help in guiding therapeutic management of PSA. The functional network analysis allowed by functional MRI is crucial to complement regional neurotransmitter deficits observed with PET. Altogether, a multimodal approach in apathy, combining PET and MRI, can allow identifying which circuits of the cortico-striato-thalamo-cortical loops are disrupted and how these circuits are modulated by other neurotransmitters.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age and younger than 75 years
* Patient with a Rankin score less then or equal to 2 and with or without apathy, demonstrated by AI scales at 3 months after stroke (apathetic patient = AI scale score > 2)
* Affiliate or beneficiary of a social security scheme
* Subjects (female study subjects and female partners of male participants) using highly effective contraceptive methods (intra-uterine device, progestin or estrogen-progestin contraceptive, sterilization)
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research)

Exclusion Criteria:

* Patients over 75 years old
* Taking of any pharmacological treatment likely to affect cholinergic systems at the time of PET-scan: Amitriptyline, Atropine, Brompheniramine, Chlorphenamine, Chlorpromazine, Clomipramine, Clozapine, Dimenhydrinate, Diphenhydramine, Doxepine, Hyoscyamine, Imipramine, Meclozine, Nortriptyline, Oxybutynine, Promethazine, Scopolamine, Trimipramine, Hydroxyzine.
* Taking of any pharmacological treatment likely to affect dopaminergic systems at the time of PET-scan: glucagon, haloperidol, reserpin
* Taking of any selective serotonine reuptake inhibitors treatment
* White matter T2 hyperintense lesions (Fazekas score > 3)
* NYHA Class III to IV Heart Failure Patient
* Patients with allergy or conter-indication to entacapone
* Subjects with positive pregnancy test (BHCG dosage and Urine dipstick), and/or currently breast-feeding
* Patients unable to come back to hospital for at least 2-follow-up visits
* Patient with a chronic neurological disorder or severe psychiatric disorder
* Patient with cognitive impairment (MoCA<24) and depression (CES-D score > 17 for men and >23 for women)
* Patient presenting a counter-indication for MRI
* Patient presenting a counter-indication for TEP with [18F]-FEOBV or [18F]-FDOPA (known allergy)
* Patient who underwent a PET examination in the previous month
* Patient with state of health not allowing a displacement in the department of imaging of the CHU: bedridden state, state of health very deteriorated
* Patient deprived of liberty by judicial or administrative decision
* Patient under legal protection or unable to express its own consent
* Subject within exclusion period from another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-04-13 (Estimated); Study Completion 2022-05-13 (Estimated)

PRIMARY OUTCOMES:
[18F]-FDOPA SUVr | Between 7 and 30 days after first visit
  Standardized uptake value for the [18F]-FDOPA radiotracer
[18F]-FEOBV SUVr | First visit (Day 0)
  Standardized uptake value for the [18F]-FEOBV radiotracer

SECONDARY OUTCOMES:
Apathy Inventory Score | First visit (Day 0)
  Apathy score from 0 to 36. Apathetic patient = score >2
Beck Anxiety Inventory (BAI) Score | First visit (Day 0)
  Beck Anxiety Inventory (BAI). Score from . Anxiety = score > 22
Lille Apathy Rating Scale (LARS) Score | First visit (Day 0)
  Complementary assessment of apathy. Score from - 36 to 36. Score < - 22 : no apathy
  * 21 to -17 : apathy tendancy
  * 16 to -10 : moderate apathy
  * 9 to 36 : severe apathy
Multidimensional Fatigue Inventory (MFI) Score | First visit (Day 0)
  The MFI contains 20 items classified into four dimensions : general fatigue, mental fatigue, reduced activities and motivation. The statements are rated on a 5-point Likert scale (from "Yes, that is true" to "No, that is not true") representing the patient's current feeling. Low MFI scores reflect a higher degree of fatigue.
Center of Epidemiology Studies Depression Scale (CES-D) Score | First visit (Day 0)
  Center of Epidemiology Studies Depression Scale (CES-D)
  The frequency of occurrence of symptoms is measured with a 4 points scale :
  o = Never
  1. = Occasionally
  2. = Quite often
  3. = Frequently The total score is between 0 and 60. Highest scores correspond to the presence of a more severe depressive symptomatology Depressive patients = score > 17 for men and >23 for women
Fractional anisotropy | First visit (Day 0)
  Fractional anisotropy measured with structural MRI
Mean diffusivity | First visit (Day 0)
  Mean diffusivity measured with structural MRI
Cerebral blood flow maps | First visit (Day 0)
  Cerebral blood flow maps provided by arterial spin labeling sequences

CONTACTS AND LOCATIONS:
Locations (1):
- Bordeaux University Hospital, Bordeaux, France